CLINICAL TRIAL: NCT03932305
Title: Randomized Controlled Trial of LUtein as a Novel Neuroprotective Adjunctive Therapy to Improve Visual Outcome of Rhegmatogenous Retinal Detachment (LUNAR Study)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Singapore National Eye Centre (Other Government)
Responsible Party: Principal Investigator, Cheung Ning, Associate Professor, Singapore Eye Research Institute
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: R1148/50/2014
Record Dates: First submitted 2019-04-18; First posted 2019-04-30 (Actual); Last update posted 2022-11-02 (Actual); Status verified 2022-10

CONDITIONS: Retinal Detachment
MeSH Terms: conditions — Retinal Detachment | interventions — Lutein

STUDY DESIGN:
Intervention Model Description: 1:1 randomisation to placebo or lutein tablets
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: double-masked for investigators and patients
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (Placebo Comparator): Patients taking inactive placebo tablets
  Interventions: Dietary Supplement: Placebo
- Lutein (Experimental): Patients taking lutein supplement
  Interventions: Dietary Supplement: Lutein

INTERVENTIONS:
Dietary Supplement: Lutein — Lutein is a common oral supplement that may have neuroprotective effect on the human retina
  Arms: Lutein
Dietary Supplement: Placebo — Inactive placebo tablet
  Arms: Control

SUMMARY:
Retinal detachment is a major cause of blindness, particularly among contemporary Asian populations due to the high prevalence of myopia. Without timely treatment, retinal detachment invariably results in blindness. As the only effective treatment is surgery, much effort has been invested to enhancing surgical outcome of retinal detachment repair. Advances in new instrumentations, viewing systems and refined surgical techniques have all contributed to improved rate of retinal re-attachment (anatomical outcome). Nevertheless, successful re-attachment of the retina after surgery does not always restore vision (visual outcome), especially when retinal detachment involves the macula ("macula-off" retinal detachment). The reason for poor visual outcome is believed to be due to apoptosis of photoreceptors, which may occur early and rapidly after the onset of retinal detachment. Neuroprotection has therefore been considered a valid strategy to improve visual outcome of retinal detachment surgery. Lutein is a promising potent neuroprotective agent for the retina, and has been shown in preliminary clinical and laboratory studies that it could salvage photorecepters in retinal detachment. We hypothesize that oral intake of lutein soon after onset of retinal detachment could prevent photoreceptor neurons from dying and thus limit the loss of vision. To test such hypothesis, we propose to conduct a double-masked, randomized controlled trial to evaluate the efficacy of lutein as an adjuvant therapy to improve visual outcome for surgical repair of primary rhematogenous retinal detachment involving the macula in Asian Singaporeans. The potential clinical and scientific significance of this trial is clear. It may provide first evidence that pharmacological neuroprotection can be used as an effective therapeutic modality in the clinical management of retinal detachment, and result in a paradigm shift in clinical practice, ultimately leading to better visual outcome and quality of life for patients undertaking surgical repair of retinal detachment.

DETAILED DESCRIPTION:
Retinal detachment is a major cause of blindness, particularly among contemporary Asian populations due to the high prevalence of myopia. Without timely treatment, retinal detachment invariably results in blindness. As the only effective treatment is surgery, much effort has been invested to enhancing surgical outcome of retinal detachment repair. Advances in new instrumentations, viewing systems and refined surgical techniques have all contributed to improved rate of retinal re-attachment (anatomical outcome). Nevertheless, successful re-attachment of the retina after surgery does not always restore vision (visual outcome), especially when retinal detachment involves the macula ("macula-off" retinal detachment). The reason for poor visual outcome is believed to be due to apoptosis of photoreceptors, which may occur early and rapidly after the onset of retinal detachment. Neuroprotection has therefore been considered a valid strategy to improve visual outcome of retinal detachment surgery. Lutein is a promising potent neuroprotective agent for the retina, and has been shown in preliminary clinical and laboratory studies that it could salvage photorecepters in retinal detachment. We hypothesize that oral intake of lutein soon after onset of retinal detachment could prevent photoreceptor neurons from dying and thus limit the loss of vision. To test such hypothesis, we propose to conduct a double-masked, randomized controlled trial to evaluate the efficacy of lutein as an adjuvant therapy to improve visual outcome for surgical repair of primary rhematogenous retinal detachment involving the macula in Asian Singaporeans. The potential clinical and scientific significance of this trial is clear. It may provide first evidence that pharmacological neuroprotection can be used as an effective therapeutic modality in the clinical management of retinal detachment, and result in a paradigm shift in clinical practice, ultimately leading to better visual outcome and quality of life for patients undertaking surgical repair of retinal detachment.

ELIGIBILITY:
Inclusion Criteria:

* Primary macula-off RRD (i.e. one that has not previously been treated with surgery)
* Able and willing to provide informed consent

Exclusion Criteria:

* Known pre-existing macular other ocular diseases (e.g., age-related macular degeneration, myopic maculopathy, diabetic macular edema, corneal diseases)
* Trauma-related RRD
* Recurrent RRD
* Macula-on RRD
* Chronic RRD (symptoms >60 days)
* History of amblyopia in the affected eye
* Known allergy to or current use of lutein supplements
* Pregnant or breastfeeding women, children (age <21 years), prisoners, cognitively impaired persons

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2016-07-25 (Actual); Primary Completion 2020-11-30 (Actual); Study Completion 2020-11-30 (Actual)

PRIMARY OUTCOMES:
Visual acuity | 6 month
  Changes in best-corrected visual acuity (BCVA) from baseline to 6-month follow-up visit

SECONDARY OUTCOMES:
Visual acuity | 12 month
  Changes in best-corrected visual acuity from baseline to 12-month follow-up visit
Retinal anatomical changes | 6 and 12 month
  Recovery of ultrastructural retinal cell layer disruptions on optical coherence tomography scans (e.g., disappearance of outer retinal disruptions at 6 and 12 month visits)
Visual function | 6 and 12 month
  Changes in visual function as measured using Pelli-Robson Contrast Sensitivity and microperimetry testing for macular function
Quality of life measures | 6 and 12 months
  Changes in "Impact of Vision Impairment Profile" based on vision impairment validated questionnaires (Lamoureux EL, Pallant JF, Pesudovs K, Rees G, Hassell JB, Keeffe JE. The impact of vision impairment questionnaire: an assessment of its domain structure using confirmatory factor analysis and rasch analysis. Invest Ophthalmol Vis Sci. 2007;48(3):1001-1006.)

IPD SHARING:
Plan to Share IPD: Undecided